CLINICAL TRIAL: NCT03001128
Title: Identification of Biomarkers to Predict Time to Plasma HIV RNA Rebound and Post-Treatment Viral Control During an Intensively Monitored Antiretroviral Pause (IMAP)
Brief Title: Biomarkers to Predict Time to Plasma HIV RNA Rebound
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5345; UM1AI068636 (NIH)
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort A: ART initiated during chronic infection: Cohort A will include 36 participants who initiated ART during chronic infection.
  Interventions: Drug: Antiretroviral treatment pause
- Cohort B: ART initiated during acute or early infection: Cohort B will include 30 participants who initiated ART during acute/early HIV infection.
  Interventions: Drug: Antiretroviral treatment pause

INTERVENTIONS:
Drug: Antiretroviral treatment pause — Antiretroviral treatment pause

SUMMARY:
The purpose of this study is to collect information about what happens when people pause, or temporarily stop taking, ART, and to collect blood samples from these people at frequent intervals. We will also study the safety of pausing ART under close observation.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies, or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally.

* Plasma HIV-1 RNA >1000 copies/mL by any assay obtained prior to initiating ART. NOTE: Documentation or candidate recall is acceptable.
* For Cohort A participants, ART initiated during chronic infection (e.g., more than 6 months after estimated date of infection, or as determined by site investigator, study team, or available medical records).
* For Cohort B, diagnosis of acute HIV infection (AHI) as defined by the criteria listed below.

Fiebig Staging Criteria (must be source documented):

* Fiebig I-II: E/CIA negative, HIV-1 RNA or p24 antigen positive, and negative or indeterminate Western blot, if performed
* Fiebig III-IV: Reactive HIV-1 antibody and negative or indeterminate results on the Western blot or Geenius HIV-1/HIV-2
* Fiebig V: Reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band NOTE A: ART must have been initiated more than 10 days after Fiebig I-II diagnosis and less than 90 days after Fiebig V diagnosis to qualify for Cohort B. NOTE B: Candidates who were diagnosed with Fiebig I-II AHI must have had a positive HIV-1 RNA test or subsequently have had a positive Western blot if no positive HIV-1 RNA test was available.

  * Receiving continuous ART for at least 2 years and on any NNRTI-, PI-, or INSTI-containing regimen.

NOTE A: ART interruptions of up to 7 days and at least 90 days prior to entry are acceptable.

NOTE B: Within- and between-class changes in ART within the previous 2 years are acceptable.

* For candidates whose ART includes an NNRTI, willingness and ability to change to a PI- or INSTI-containing regimen for at least 4 weeks prior to ART interruption and the local availability of such a regimen.
* Nadir CD4+ cell count ≥200 cells/mm3.

NOTE: Candidate recall or documentation is acceptable.

* CD4+ cell count ≥500 cells/mm3 obtained within 90 days prior to study entry in a US laboratory that has is compliant with Clinical Laboratory Improvement Amendments (CLIA) or its equivalent or in any network approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance (EQA) programs.
* One documented plasma HIV-1 RNA that is below the limit of detection of an FDA-approved assays (limit of detection: 75, 50, 40, or 20 copies/mL) between 12 and 24 months prior to the screening HIV-1 RNA and one documented HIV-1 RNA that is below the limit of detection of the FDA-approved assays (limit of detection: 75, 50, 40, or 20 copies/mL) collected fewer than 12 months prior to the screening HIV-1 RNA.
* Plasma HIV-1 RNA level below the limit of assay quantification within 90 days prior to entry.
* The following laboratory values obtained within 90 days prior to entry by any US laboratory that is compliant with CLIA or its equivalent or in any network approved non-US laboratory that operates in accordance with GCLP and participates in appropriate EQA programs.

Absolute neutrophil count (ANC) ≥750 cells/mm3 Hemoglobin ≥11.0 g/dL for men and ≥10.0 g/dL for women Platelet count ≥100,000/mm3 Creatinine ≤1.5 mg/dL Aspartate aminotransferase (AST) (SGOT) ≤1.5x upper limit of normal (ULN) Alanine aminotransferase (ALT) (SGPT) ≤1.5x ULN

* HCV antibody negative result obtained within 90 days prior to study entry or, if the HCV antibody result is positive, a negative HCV RNA result within 90 days prior to study entry and no positive HCV RNA result within 24 weeks prior to entry.
* Ability and willingness of participant to provide informed consent.
* Willingness to have blood samples collected and stored indefinitely and used for HIV-related research purposes.
* For females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy and/or bilateral salpingectomy), a negative serum or urine pregnancy test within 48 hours prior to study entry by any clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care CLIA-waived test, or at any network approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practices and participates in appropriate external quality assurance programs.

NOTE: Acceptable documentation of hysterectomy and bilateral oophorectomy, bilateral salpingectomy, tubal micro-inserts, partner who has undergone vasectomy, and menopause is participant-reported history.

* All participants must agree to use barrier protection (e.g., condoms, dental dams) for all sexual activity throughout the entire course of the study to prevent HIV transmission.
* All participants must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, or in vitro fertilization). If participating in sexual activity that could lead to pregnancy, the participant/partner must use at least two reliable forms of contraceptives (e.g., condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; hormone-based contraception), with at least one being a barrier method, during the study.
* Site investigator anticipates that a fully active alternative ART regimen could be constructed and would be available in the event of virologic failure on the participant's current ART regimen.
* Absence of either active hepatitis B virus (HBV) infection, indicated by a negative hepatitis B surface antigen (HBsAg) or HBV viral load assays within 90 days prior to entry or known chronic hepatitis B infection based on a previously positive HBV DNA or positive HBsAg without a subsequent positive hepatitis B surface antibody (HBsAb).

Step 1 Exclusion Criteria:

* Any plasma HIV-1 RNA at or above the limit of detection of the FDA-approved assays (limit of detection: 75, 50, 40, or 20 copies/mL) within 24 months prior to entry.

NOTE: A single unconfirmed "blip" (i.e., plasma HIV-1 RNA over limit of detection but <200 copies/mL) is allowed if preceded and followed by values below the limit of detection and if the blip occurred more than 6 months prior to study entry.

* Currently breastfeeding or plans on breastfeeding during the course of the study or is pregnant.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.
* Any history of an AIDS-defining illness using the current list on the U.S. Centers for Disease Control and Prevention (CDC)'s website.
* Receipt of any study-defined prohibited medications within 6 months prior to entry.
* Prior history of difficulty establishing venous access or current contraindication for leukapheresis, in the opinion of the site investigator and based on assessments.
* Receipt of any vaccination within 1 week prior to entry.

NOTE: The entry visit must be scheduled to ensure that 1 week has elapsed after any vaccination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected men and women ≥18 to ≤70 years of age, maintained on suppressive ART for a minimum of 2 years with CD4+ count ≥500 cells/mm3 and nadir CD4+ count ≥200 cells/mm3.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Time from ART discontinuation to HIV RNA rebound | Up to 96 weeks following ART discontinuation
  Time from ART discontinuation (start of MAP) to HIV RNA rebound to ≥ 1,000 copies/mL
Frequency of sustained post-treatment HIV control | ≥24 weeks off ART without meeting ART re-initiation criteria
  Frequency of sustained post-treatment HIV control in participants treated during early and chronic infection undergoing an IMAP
Association between pre-IMAP CA-RNA and time to HIV rebound | Up to 96 weeks following ART discontinuation
  Association between pre-IMAP CA-RNA and time to HIV rebound

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Li, MD, MMS, Study Chair — Brigham and Women's Hospital ACTG CRS; David Smith, MD, MAS, Study Chair — University of California San Diego AVRC CRS
Locations (18):
- United States (16):
  - 601 University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - 701 University of California, San Diego AntiViral Research Center CRS, San Diego, California
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - 2701 Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - 101 Massachusetts General Hospital (MGH) CRS, Boston, Massachusetts
  - 107 Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - 3201 Chapel Hill CRS, Chapel Hill, North Carolina
  - 3203 Greensboro CRS, Greensboro, North Carolina
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - 3652 Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - 31443 Trinity Health and Wellness Center CRS, Dallas, Texas
- 5401 Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, PR, Puerto Rico
- 31802 Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok, Patumwan, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gianella S, Yu T, Wang R, Ignacio C, Schanz M, Kouyos RD, Caballero G, Gaitan NC, Rawlings S, Kuster H, Metzner KJ, Gandhi RT, Li JZ, Gunthard HF, Smith DM, Chaillon A. Viral and Immune Risk Factors of HIV Rebound After Interruption of Antiretroviral Therapy. J Infect Dis. 2025 Jun 2;231(5):1221-1229. doi: 10.1093/infdis/jiae585. PMID 39661441
- [Derived] Li JZ, Melberg M, Kittilson A, Abdel-Mohsen M, Li Y, Aga E, Bosch RJ, Wonderlich ER, Kinslow J, Giron LB, Di Germanio C, Pilkinton M, MacLaren L, Keefer M, Fox L, Barr L, Acosta E, Ananworanich J, Coombs R, Mellors J, Deeks S, Gandhi RT, Busch M, Landay A, Macatangay B, Smith DM; AIDS Clinical Trials Group A5345 Study Team. Predictors of HIV rebound differ by timing of antiretroviral therapy initiation. JCI Insight. 2024 Feb 8;9(3):e173864. doi: 10.1172/jci.insight.173864. PMID 38329130
- [Derived] Dube K, Eskaf S, Barr L, Palm D, Hogg E, Simoni JM, Sugarman J, Brown B, Sauceda JA, Henley L, Deeks S, Fox L, Gandhi RT, Smith D, Li JZ. Participant Perspectives and Experiences Following an Intensively Monitored Antiretroviral Pause in the United States: Results from the AIDS Clinical Trials Group A5345 Biomarker Study. AIDS Res Hum Retroviruses. 2022 Jun;38(6):510-517. doi: 10.1089/AID.2021.0170. Epub 2022 Apr 21. PMID 35323030
- [Derived] Diepstra KL, Barr L, Palm D, Hogg E, Mollan KR, Henley L, Stover AM, Simoni JM, Sugarman J, Brown B, Sauceda JA, Deeks S, Fox L, Gandhi RT, Smith D, Li JZ, Dube K. Participant Perspectives and Experiences Entering an Intensively Monitored Antiretroviral Pause: Results from the AIDS Clinical Trials Group A5345 Biomarker Study. AIDS Res Hum Retroviruses. 2021 Jun;37(6):489-501. doi: 10.1089/AID.2020.0222. Epub 2021 Feb 16. PMID 33472545